CLINICAL TRIAL: NCT06238544
Title: An Open Label, Multicenter Study to Evaluate the Long-term Safety and Tolerability of HRS-5965 in Patients With Paroxysmal Nocturnal Hemoglobinuria
Brief Title: Long-term Safety and Tolerability of HRS-5965 in Patients With Paroxysmal Nocturnal Hemoglobinuria
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chengdu Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-5965-203
Record Dates: First submitted 2024-01-22; First posted 2024-02-02 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRS-5965 Group (Experimental)
  Interventions: Drug: HRS-5965 tablets; Drug: HRS-5965 Capsules

INTERVENTIONS:
Drug: HRS-5965 tablets — HRS-5965 tablets until the end of study treatment
Drug: HRS-5965 Capsules — HRS-5965 capsules.

SUMMARY:
This is a multicenter, single-arm, open-label study. Patients with Paroxysmal Nocturnal Hemoglobinuria who had previously received and completed the HRS-5965 study well included. All eligible subjects received HRS-5965 tablets or capsules until the end of treatment in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have previously received and completed HRS-5965 study treatment, and are judged by the investigator to have treatment benefit and may benefit from continued treatment of HRS-5965 and patients in the control group of who received eculizumab treatment.

Exclusion Criteria:

1. Known or suspected hereditary or acquired complement deficiency;
2. History of infection with capsular bacteria (e.g., meningococcus, pneumococcus, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2024-02-06 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events. | Every six months,for about 3 years

SECONDARY OUTCOMES:
Proportion of participants achieving sustained hemoglobin levels ≥ 12 g/dL in the absence of red blood cell transfusions was assessed every half a year during treatment.. | Every six months ,for about 3 years
Proportion of participants who remain free from transfusions was assessed every half a year during treatment.. | Every six months,for about 3 years
Rate of breakthrough hemolysis was assessed every half a year during treatment | Every six months,for about 3 years
Proportion of participants with Major Adverse Vascular Events MAVEs. | Every six months,for about 3 years
Plasma concentration of HRS-5965. | Start of Treatment to end of study，for about 3 years

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - The Blood Disease Hospital of the Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Undecided